CLINICAL TRIAL: NCT04444622
Title: Phase IIB Open-Label Study to Assess the Safety and Efficacy of STIMVAX® as Third-line Therapy for Metastatic Colorectal Cancer
Brief Title: Immunotherapy for Third Line Metastatic Colorectal Cancer
Acronym: STIMVAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-032-MCRC3-STIM
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: immunotherapy; cancer vaccine; colorectal cancer; AlloStim; MSI-S
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AlloStim (Experimental): AlloStim is administered in three cycles:
  Cycle 1 Day 0: 0.5ml ID AlloStim® Day 7: 0.5ml ID AlloStim® Day 14: 0.5ml ID AlloStim® Day 21: 0.5ml ID AlloStim® Day 28: 0.5ml ID AlloStim®
  Cycle 2 Day 42: 0.5ml ID AlloStim® Day 49: 0.5ml ID AlloStim® Day 56: 0.5ml ID AlloStim® Day 63: 0.5ml ID AlloStim® Day 70: 0.5ml ID AlloStim® + 3ml IV AlloStim®
  Cycle 3 Day 84: 0.5ml ID AlloStim® Day 91: 0.5ml ID AlloStim® Day 98: 0.5ml ID AlloStim® Day 105: 0.5ml ID AlloStim® Day 112: 0.5ml ID AlloStim® + 3ml IV AlloStim®
  Interventions: Biological: AlloStim

INTERVENTIONS:
Biological: AlloStim — Living bioengineered, non-genetically manipulated, activated Th1-like immune cells differentiated and expanded from precursor cells purified from blood of healthy unrelated donors
  Other Names: StimVax

SUMMARY:
This is a Phase IIB multi-site, open label study of a next generation immunotherapy for third-line MSI-S metastatic colorectal cancer using an "off-the-shelf", non-genetically manipulated living immune cell product (AlloStim) derived from the blood of healthy donors.

DETAILED DESCRIPTION:
This is a Phase IIB open label immunotherapy protocol called "StimVax". The protocol design is based upon information obtained from a previous Phase IIA dose level and dose frequency ranging study. The population targeted is MSI-S metastatic colorectal cancer previously treated with two lines of chemotherapy regimens, one containing oxaliplatin and the other containing irinotecan. This population is not considered to be responsive to immunotherapy.

The study drug is called "AlloStim". AlloStim is an "off-the-shelf", non-genetically-manipulated, living immune cell immunotherapy. AlloStim is derived from precursors purified from the blood of healthy donors and grown and differentiated in specialized bioreactors in the laboratory. Because the donors are intentionally mis-matched to the host, AlloStim is completely eliminated by the host in a non-toxic rejection response within 24h of administration.

Unlike autologous immune cell therapies, like CAR-T cells or TIL cells, AlloStim is allogeneic and is not intended to directly kill tumors. Rather, the novel AlloStim mechanism is designed to modify and train the host immune system to kill tumors and prevent tumor growth and spread. Uniquely, the AlloStim mechanism is also designed to increase Th1/Th2 balance, activate innate effector cells (such as NK and NKT), counter-regulate the immune suppressive and immune evasion mechanisms that tumors use to evade immune elimination both systemically and in the tumor microenvironment.

The AlloStim mechanism creates self-amplifying waves of temporal and spatial immune effects that can lead to an initial non-specific cellular innate NK cell immune response followed by a tumor-specific killer T-cell immune response specific for the host tumor through a combination of immune processes called "allo-priming" and "in-situ vaccination".

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and female subjects aged 18-80 years at screening visit
2. Pathologically confirmed diagnosis of colorectal adenocarcinoma
3. Presenting with metastatic disease:
4. Previous treatment failure of two previous lines of active systemic chemotherapy:

   * Previous chemotherapy must have included an oxaliplatin-containing (e.g. FOLFOX) and an irinotecan-containing (e.g. FOLFIRI) regimen
   * With or without bevacizumab
   * Administered in adjuvant setting or for treatment of metastatic disease
   * If KRAS wild type, must have at least one prior anti-EGFR therapy
   * Treatment failure can be due to disease progression or toxicity
   * Disease progression on second line therapy must be documented radiologically and must have occurred during or within 30 days following the last administration of treatment for metastatic disease
5. ECOG performance score: 0-1
6. Adequate hematological function:

   * Absolute granulocyte count ≥ 1,200/mm3
   * Platelet count ≥ 100,000/mm3
   * PT/INR ≤ 1.5 or correctable to <1.5 at time of interventional procedures
   * Hemoglobin ≥ 9 g/dL (may be corrected by transfusion)
7. Adequate Organ Function:

   * Creatinine ≤ 1.5 mg/dL
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Alkaline phosphatase ≤ 2.5 times ULN *
   * Aspartate aminotransferase (AST) or (SGOT) ≤ 2.5 times ULN *
   * Alanine aminotransferase (ALT) or (SGPT) ≤ 2.5 times ULN * *or ≤5x ULN if liver involvement
8. EKG without clinically relevant abnormalities
9. Female subjects: Not pregnant or lactating
10. Patients with child bearing potential must agree to use adequate contraception
11. Study specific informed consent in the native language of the subject.

Exclusion Criteria:

1. high frequency microsatellite instability (MSI-H)
2. Bowel obstruction or high risk for obstruction if tumors become inflamed
3. Moderate or severe ascites requiring medical intervention
4. Clinical evidence or radiological evidence of brain metastasis or leptomeningeal involvement
5. Peritoneal carcinomatosis
6. Symptomatic asthma or COPD
7. Pulmonary lymphangitis or symptomatic pleural effusion (grade ≥ 2) that results in pulmonary dysfunction requiring active treatment; or, oxygen saturation <92% on room air
8. Bevacizumab (Avastin®) treatment within 6 weeks of baseline scheduled biopsy procedure
9. Any of the following mood disorders: active major depressive episode, history of suicidal attempt or ideation
10. Prior allogeneic bone marrow/stem cell or solid organ transplant
11. Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 5 mg/day of prednisone) within 30 days of the first day of study drug treatment

    * Topical corticosteroids are permitted
12. Prior diagnosis of an active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis).

    * Well controlled Type I diabetes allowed
13. Prior experimental therapy
14. History of blood transfusion reactions
15. Progressive viral or bacterial infection

    * All infections must be resolved and the subject must remain afebrile for seven days without antibiotics prior to being placed on study
16. Cardiac disease of symptomatic nature
17. History of HIV positivity or AIDS
18. Concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless such medications can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to biopsy procedures
19. History of severe hypersensitivity to monoclonal antibody drugs
20. Psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation.
21. Subjects that lack ability to provide consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | date of death from any cause, whichever came first, assessed up to 12 months from accrual
  measurement of the survival on experimental treatment
Incidents of Adverse Events (AE) | day 0 to 1 year
  to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mt. Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Summit Health, Florham Park, New Jersey
  - Hirschfield Oncology Center, The Bronx, New York

REFERENCES:
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441